CLINICAL TRIAL: NCT06686056
Title: A Single-Center, Open-Label, Randomized, Parallel Controlled Trial Evaluating the Effectiveness of Artificial Intelligence-Enhanced Management for Coronary Heart Disease (AIM-CHD) Delivered Via Mobile Application
Brief Title: Artificial Intelligence-Enhanced Management for Coronary Heart Disease (AIM-CHD) : Impact on Cholesterol and Other CHD Risk Factors
Acronym: AIM-CHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-GSP-GG-4
Record Dates: First submitted 2024-11-11; First posted 2024-11-13 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Secondary Prevention of Coronary Heart Disease
Keywords: Coronary heart disease; secondary prevention; mobile health; artificial intelligence
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AIM-CHD Mobile Health Intervention Group (Experimental): Participants in the intervention group will be trained to use the AIM-CHD for post-discharge care，while also receiving post-discharge usual care.
  Interventions: Combination Product: AIM-CHD Mobile Health Intervention; Combination Product: Usual post-discharge care
- Standard Post-Discharge Care Group (Active Comparator): Participants in the control group will receive usual post-discharge care, which includes oral and written instructions on sustained pharmacotherapy regimens, recommended follow-up frequency, and lifestyle modifications.
  Interventions: Combination Product: Usual post-discharge care

INTERVENTIONS:
Combination Product: AIM-CHD Mobile Health Intervention — The AIM-CHD platform synchronizes data from hospitalization records, questionnaires, AI-powered voice follow-ups, and wearable devices to perform risk stratification and manage uncontrolled risk factors. It provides individualized follow-up plans, medication reminders, and lifestyle education, with real-time assessments of vital health metrics to prompt necessary in-person consultations. The app offers online consultation access and emergency services through Fuwai Hospital. Additionally, it delivers personalized patient education, aligning with the latest clinical guidelines.
  Arms: AIM-CHD Mobile Health Intervention Group
Combination Product: Usual post-discharge care — Usual post-discharge care includes oral and written instructions on sustained pharmacotherapy regimens, recommended follow-up frequency, and lifestyle modifications.

SUMMARY:
The goal of this clinical trial is to find out if an artificial intelligence (AI)-enhanced mobile app can help people with coronary heart disease (CHD) better manage their health after being discharged from the hospital. The main questions it aims to answer are:

1. Does the AI-enhanced app help lower bad cholesterol (LDL-C) levels within 3 months after leaving the hospital?
2. Does the app improve other health measures, like blood pressure, blood sugar control, weight, medication adherence and cardiac events?

Researchers will compare the AI-enhanced app to usual care, where participants receive usual health advice without using the app.

Participants will:

1. Be randomly assigned to use either the AI-enhanced app or receive usual care.
2. Use the app to track and manage their health, receive reminders, and get educational tips.
3. Attend checkups at 3 months to measure cholesterol levels and other health outcomes.

The study hopes to show that using an AI-enhanced app can make it easier for people with CHD to stay healthy and avoid future heart problems.

DETAILED DESCRIPTION:
The AIM-CHD app was developed by a diverse team at Fuwai Hospital, including doctors, nurses, patients, and software engineers. It gathers information from synchronized hospital records, questionnaires, intelligent voice follow-ups, and wearable devices. Using this data, it categorizes patients by risk level, detects unmanaged risk factors, and generates individualized follow-up schedules and intervention plans. When risk factors are not well controlled, the app alerts patients to these issues. It also reminds users to monitor their health markers regularly, follow prescribed medication routines, and offers personalized health education focused on lifestyle adjustments. The app can assess the severity of blood pressure, heart rate, blood glucose, and lipid levels, advising patients to seek in-person consultations if necessary. AIM-CHD also recognizes emergency scenarios and provides options for online consultations or immediate help from Fuwai Hospital to prevent treatment delays. The platform leverages artificial intelligence (AI) for efficient lab report image recognition and speech-to-text conversion, streamlining follow-up care. Additionally, it offers customized patient education. The AIM-CHD's intervention goals and strategies are grounded in the latest clinical guidelines. The system is built with a front-end and back-end separation architecture: the back-end is developed with the .NET framework using C#, while the front-end is a WeChat mini-program created with JavaScript and React.

ELIGIBILITY:
Inclusion Criteria:

* CHD patients aged 18-85 years
* ability of the patient or close relatives to use smartphones and applications
* willingness to participate and sign the informed consent form

Exclusion Criteria:

* severe cognitive impairment
* advanced malignant tumors
* expected survival of less than 3 months
* severe multi-organ failure
* refusal to sign the informed consent form

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Actual)
Dates: Start 2024-11-23 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
LDL-C levels | measured at 3 months post-discharge.
  LDL-C levels (mmol/L)

SECONDARY OUTCOMES:
LDL-C Target Attainment Rate | assessed at 3 months post-discharge
  Proportion of patients achieving LDL-C <1.8 mmol/L
Blood Pressure Control Rate | assessed at 3 months post-discharge
  Proportion of patients with controlled blood pressure, defined as systolic pressure <130 mmHg and diastolic pressure <80 mmHg.
Glycosylated Hemoglobin Levels | assessed at 3 months post-discharge
Smoking Rate | assessed at 3 months post-discharge
  Proportion of patients who are still smoking
BMI | assessed at 3 months post-discharge
  body mass index
Cardiovascular Composite Endpoint Events | assessed at 3 months post-discharge
  Incidence of all-cause mortality, non-fatal myocardial infarction, stroke, and rehospitalization.
Medication Adherence | assessed at 3 months post-discharge
  Proportion of patients adhering to antiplatelet agents and statins, defined as taking medications for more than 80% of the prescribed time over the past month.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Sciences/National Center for Cardiovascular Diseases, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The individual participant data collected in this study contains sensitive information. Although de-identified, the data will not be publicly shared to protect participant privacy and in accordance with the requirements of the ethics committee.

REFERENCES:
- [Derived] Ba Z, Zhao S, Liu M, Chen G, Lian X, Yu F, Su Y, Wang Z, Yang L, Wang X, Zhang X, Yuan J, Gao X, Zhao W, Wu Y. Effectiveness of an AI-enhanced management system for coronary heart disease (AIM-CHD): rationale and design of a single-centre, open-label, randomised, parallel-controlled trial. BMJ Open. 2025 Sep 14;15(9):e105597. doi: 10.1136/bmjopen-2025-105597. PMID 40953879